CLINICAL TRIAL: NCT03936153
Title: An Open-label, Single-arm, Multi-center Phase 2 Study to Evaluate the Efficacy and Safety of Abexinostat as Monotherapy in Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Study to Evaluate Efficacy and Safety of Oral Abexinostat in Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xynomic Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYN-606
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Diffuse Large B-cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — abexinostat

STUDY DESIGN:
Intervention Model Description: A single arm treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abexinostat 80 mg bis in die (BID) (Experimental): Abexinostat 80 mg BID
  Interventions: Drug: abexinostat

INTERVENTIONS:
Drug: abexinostat — abexinostat tablet

SUMMARY:
An open-label, single-arm, multi-center phase 2 study to evaluate the efficacy and safety of abexinostat, as monotherapy in patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL)

DETAILED DESCRIPTION:
An open-label, single-arm, multi-center phase 2 study to evaluate the efficacy and safety of oral histone deacetylase (HDAC)-inhibitor abexinostat, as monotherapy in patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL)

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diffuse large B-cell lymphoma (DLBCL);
2. Have received only two prior standard therapy lines for diffuse large B-cell lymphoma (DLBCL) including anti- cluster of differentiation antigen (anti-CD20) antibody and cytotoxic therapy;
3. Confirmed to be unresponsive to the last line of therapy, or have disease progression following the last line of therapy;
4. Have at least one radiologically measurable lymph node or extranodal lymphoid malignant lesion;
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2;
6. Meet various hematological, liver and renal function lab parameters.

Exclusion Criteria:

1. Have primary central nervous system (CNS) lymphoma or secondary central nervous system (CNS) infiltration, transformed lymphoma, unclassified B-cell lymphoma with features intermediate between DLBCL and classical Hodgkin's lymphoma (HL), primary effusion lymphoma, plasma lymphoma;
2. Toxicity not yet recovered from previous anti-tumor therapies;
3. Uncontrolled systemic infections or infections requiring intravenous antibiotics;
4. Have received steroid hormone, chemotherapy, targeted therapy, radiotherapy, antibody-based therapies, within a specified amount of time per protocol;
5. Unable to swallow tablets, or presence of significant functional gastrointestinal disorders that may affect the intake, transport or absorption of the study drug;
6. Have received autologous stem cell transplant,or allogeneic stem cell transplant within a certain amount of time as specified in protocol;
7. Presence of active graft-versus-host reaction;
8. Have undergone a major surgery within the last month;
9. Evidence of possible human immunodeficiency virus (HIV) infection or hepatitis C virus (HCV) infection;
10. Have any cardiac impairment as defined per protocol;
11. Have prior history of malignancies other than diffuse large B-cell lymphoma (DLBCL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Clinical effect by evaluating the objective response rate (ORR) | up to 56 days
  To evaluate the objective response rate (ORR) of abexinostat in patients with relapsed/refractory diffuse large B-cell lymphoma (DLBCL) as assessed by an independent central imaging review.

SECONDARY OUTCOMES:
Objective Response | up to 56 days
  Objective response rate (ORR) as assessed by the investigator
Progression-free survival | Up to 2 years
  Progression-free survival (PFS), defined as the time from the initiation of treatment to disease progression or death as assessed by the independent Central Imaging Review and the Investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai SHI, Prof, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (23):
- China (23):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliate Hospital of Dalian Medical University, Dalian
  - Fujian Medical University Union Hospital, Fuzhou
  - Fujian Provincial Cancer Hospital, Fuzhou
  - Cancer Center of Guangzhou Medical University, Guangzhou
  - Sun Yai-Sen Memorial Hospital, Sun Yai-Sen University, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - The Affiliated Tumor Hospital of Harbin Medical University, Harbin
  - The First Hospital of Lanzhou University, Lanzhou
  - Linyi Cancer Hospital, Linyi
  - Nantong Tumor Hospital, Nantong
  - Shanghai Jiao Tong University School Medicine, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Second People's Hospital of Shenzhen, Shenzhen
  - The Forth Hospital of Hebei Medical University, Shijiazhuang
  - First Hospital of Shanxi Medical University, Taiyuan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No